CLINICAL TRIAL: NCT06453473
Title: The Transfer Effects of Stationary Bicycle Perturbation Training on Older Adults' Cycling Skills and Behavior (BiPerAge): a Single Blind Randomized Controlled Trial
Brief Title: Transfer Effects of Stationary Bicycle Perturbation Training on Older Adults' Cycling Skills
Acronym: BiPerAge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BGU-IBA-2024-BiPerAge
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Older Adults; Exercise Training; Bicycling
Keywords: Bicycling; Perturbation; Balance control; Falls

STUDY DESIGN:
Intervention Model Description: BiPerAge is a parallel group (1:1), randomized controlled trial with a duration of 3 years and a recruitment period between September 2024 and December 2025.
  Baseline data collection (T0) takes place in-person in the study center and in the cycle course on two different days within approximately 14 days. Except for cognitive function, same data are collected of all participants after the 3 months intervention period (T1), regardless of their compliance. In addition, participants will be followed up 6-9 months after T1 (T2) related to seasonal time frames (after winter season).
Who Masked: Outcomes Assessor
Masking Description: Outcome measures will be obtained by two research assistants in each country who are blinded to group allocation. Participants will not fully be blinded to group allocation since they notice whether perturbation occur during training. However, both groups will be told that the primary aim of the study is to improve cycling skills by training on an indoor, stationary bicycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- training on the PerStBiRo with pertubation (PerTSBR) (Experimental): The experimental group will pedall on the PerStBiRo system like the active comparator group but will receive additional roll- and pitch-angles balance perturbations.
  Interventions: Other: TSBR; Other: PerTSBR
- unperturbed training on the PerStBiRo (TSBR) (Active Comparator): The active comparator group will pedall on the PerStBiRo system without perturbations.
  Interventions: Other: TSBR

INTERVENTIONS:
Other: TSBR — The intervention consists of 20 training sessions on the PerStBiRo system (~ twice a week within 3 months period). Each session lasts for 20 minutes and includes three parts: stage 1) warm up, stage 2) main exercise and stage 3) cool down.
  Stage 1 contains 3 minutes of self-paced pedalling with the same bicycle resistance. At Stage 2, the main exercise, all participants will perform a 15-minute hands-free cycling training on the PerStBiRo system with a pulse watch to maintain moderate-intensity training, corresponding to 64-76% of the predicted maximal heart rate (Borg scale 12-14), including cognitive tasks projected at a screen in front of the participant. Stage 3 includes the cool down with 2 minutes of self-paced pedalling without bicycle resistance and cognitive tasks. During the training sessions, all participants will wear a loose safety harness that can arrest falling using the PerStBiRo system, but still allow comfortable pedalling.
Other: PerTSBR — Participants of the intervention group will receive a combination of lateral and medial tilting unannounced perturbations during stage 2 of the TSBR training. This will be provided by roll and pitch angles (tilt) balance perturbations that aim to evoke trunk and arm balance recovery responses.
  Arms: training on the PerStBiRo with pertubation (PerTSBR)

SUMMARY:
The Israeli research group of this trial has developed the Perturbation Stationary Bicycle Robotics (PerStBiRo) system that can challenge balance while sitting. With this system, unexpected perturbations can be provided under controlled and safe conditions. Within the BiPerAge-project it will be evaluated if 20 training sessions (20 minutes each) on the PerStBiRo system will lead to transfer effects on safe cycling skills of community-dwelling older adults (age 65 years and older). The ability to cycle safely will be tested prior and after the training period using a cycling course, which consists of variant tasks requiring motor and cognitive skills.

DETAILED DESCRIPTION:
Cycling is a form of physical activity that is positively associated with health and functional benefits. However, there is a significant association between increased bicycle use and bicycle accidents with higher risks of severe injuries especially for older adults. This could be partly explained by deterioration of the balance control during aging. On the one hand, training of balance-challenging situations in daily traffic situation is hardly possible under "real-world" conditions for safety reasons. On the other hand, the use of a stationary bicycle alone has not been shown to specifically train balance skills and cycling competence. To overcome this issue the Israeli research group of this trial has developed the Perturbation Stationary Bicycle Robotics (PerStBiRo) system that can challenge balance while riding in a controlled and safe condition.

The main and overarching objective of our proposed project is to investigate transfer effects of a training on the PerStBiRo system with perturbation (PerTSBR - intervention group) on cycling competence of community-dwelling older adults (age 65 years and older) in comparison to a training on the same system without perturbation (TSBR - active control group). The cycling competence as our primary outcome will be measured by a standardized cycle course before and after the 3 months intervention period. The cycle course, which is validated in a recent study (SiFAr) of our research group, consists of various tasks requiring motor and cognitive skills related to traffic situations in daily life.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide informed consent and accept randomization to either study arm
* Ability to come to cycle course testing locations
* ≥3 errors in pre-test of cycle course

Exclusion Criteria:

* Severe diseases e.g. ischemic heart disease which restricts exercise, chronic obstructive pulmonary disease (COPD), uncontrolled blood pressure, manifest osteoporosis or any other disease leading to increased fracture risks
* A period less than one year after hip or knee replacement surgery or after fractures of the lower extremities
* Amputation of a lower limb
* Neurological diseases or 6-month after a stroke
* Inability to ambulate independently
* Severe visual impairments (blindness), non-compensable hearing
* Cognitive impairment, scoring less than 24 on the MMSE (Mini-Mental State Examination), inability to understand and follow instructions
* Participation in another intervention trial at the same time or within the previous 6 months

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of faults in the cycling course | changes over a period of 3 months and after a follow-up period of 6-9 months
  The cycling competence will be tested in a standardized cycling course, including the following tasks: slalom, slow cycling within a marked lane, dismounting into a marked zone, getting on the bike, cycling through a narrow alley, turning to the off-side, braking with pinpoint accuracy. Mean change of number of faults in the cycling course will be tested between pre- and postintervention.

SECONDARY OUTCOMES:
Balance Error Scoring System (BESS) | changes over a period of 3 months and after a follow-up period of 6-9 months
  mean change in sumscore counting the errors, or deviations from the proper stance (0-30 error points) for measurement of static balance, higher error points indicate worse balance
5 Chair Stand Test | changes over a period of 3 months and after a follow-up period of 6-9 months
  mean change of time in seconds for measurement of muscle power of the legs
Four Square Step Test | changes over a period of 3 months and after a follow-up period of 6-9 months
  mean change of time in seconds for measurement of dynamic balance

OTHER OUTCOMES:
Bicycle falls efficacy scale | changes over a period of 3 months and after a follow-up period of 6-9 months
  mean change of sumscore in an own developed questionnaire regarding concerns about falling from the bicycle (14-56 points), higher score indicates increased concerns about falling off the bicycle
Short Physical Performance Battery (SPPB) | changes over a period of 3 months and after a follow-up period of 6-9 months
  mean change in sumscore (0-12 points) for measurement of static balance, gait speed and chair stand test, more points indicate better physical functioning
Heart rate variability (HRV) | changes over a period of 3 months and after a follow-up period of 6-9 months
  mean change of measured heart rate variability , higher scores indicate better cardiac autonomic nervous system function
Balance recovery score | changes over a period of 3 months and after a follow-up period of 6-9 months
  mean change of measured balance recovery score that is based on the time needed to counteract the perturbations on the stationary bike during a standardized perturbation intervention, higher scores indicate better balance reactions
Predicted maximal oxygen consumption (VO₂max) | changes over a period of 3 months and after a follow-up period of 6-9 months
  mean change of predicted maximal oxygen consumption estimated via the submaximal Ekblom-Bak cycle ergometer test, higher maximal oxygen consumption indicates better physical fitness

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kob, PhD, Principal Investigator — Institute for Biomedicine of Aging, Friederich-Alexander-Universität Erlangen-Nürnberg
Locations (2):
- Friedrich-Alexander-Universität Erlangen-Nürnberg, Institut für Biomedizin des Alterns, Nuremberg, Bavaria, Germany
- Physical Therapy department, faculty of health sciences, Ben-Gurion University of the Negev, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: Yes
Data relative to this work will be available upon reasonable request to the principal investigators.
Supporting Information: Study Protocol, ICF
Time Frame: The data could be requested after the publication of the primary study results and will be kept available for at least 10 years after completion of the study.
Access Criteria: Data relative to this work will be available upon reasonable request to the principal investigators.